CLINICAL TRIAL: NCT07097077
Title: Study of Functional Magnetic Resonance Signal Variations in Patients Undergoing Anterior Cruciate Ligament Reconstruction With the Application of a Dedicated Neuromotor Training
Acronym: ACL-fMRI-TNMT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stefano Zaffagnini (Other)
Collaborators: IRCCS Istituto delle Scienze Neurologiche di Bologna (Other); ISOKINETIC ER SRL (Unknown)
Responsible Party: Sponsor-Investigator, Stefano Zaffagnini, Full Professor Medicine and Surgery, University of Bologna, Istituto Ortopedico Rizzoli
Organization: Istituto Ortopedico Rizzoli (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACL-fMRI-TNMT
Record Dates: First submitted 2025-07-11; First posted 2025-07-31 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: fMRI; ACL Injury; Rehabilitation Exercise; Neuromuscular Control
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ACL Patients performing neuromotor training (Experimental)
  Interventions: Other: Effect of targeted neuromotor training in patients undergoing ACL reconstruction on the volumetric activation of cerebral cortex regions during fMRI.

INTERVENTIONS:
Other: Effect of targeted neuromotor training in patients undergoing ACL reconstruction on the volumetric activation of cerebral cortex regions during fMRI. — The effect of targeted neuromotor training in patients undergoing ACL reconstruction on the volumetric activation of cerebral cortex regions during fMRI. Differences in brain activation will be assessed between timepoint t0 (after ACL reconstruction surgery and before the start of training) and timepoint t1 (after completion of the training).

SUMMARY:
Lower limb injuries represent the majority of sports-related injuries, with knee injuries being among the most common. In particular, anterior cruciate ligament (ACL) injuries are considered highly devastating and career-threatening for both professional and amateur athletes. Current surgical and rehabilitation treatments often fail to provide fully satisfactory short- and long-term outcomes. A very high risk of re-injury exists, especially in younger patients, with up to 35% experiencing a second ACL injury, alongside a significant long-term risk of early knee osteoarthritis.

Most ACL injuries are non-contact or indirect contact injuries, implicating biomechanical factors and neuromuscular control as key determinants of injury mechanisms. Recent literature shows that patients suffering a non-contact ACL injury have a higher risk of re-injury compared to those with contact injuries, suggesting a significant cognitive component in injury processing, surgery, rehabilitation, and return to sport.

Recent rehabilitation studies have introduced targeted neuromotor training designed to "rebuild" biomechanical and neuromuscular patterns to avoid mechanisms leading to re-injury. Movement quality tests are used post-training to confirm the reduction of risky biomechanical patterns, often resulting in a score indicating movement quality.

Given the brain's involvement in such injuries, pioneering studies have used functional magnetic resonance imaging (fMRI) to investigate changes in cortical brain areas following ACL injury and reconstruction. Evidence shows adaptations in both central and peripheral nervous systems, with altered sensorimotor cortex activation in patients during simple motor tasks, differing from healthy subjects. Prefrontal cortex alterations correlate with severe quadriceps muscle activation asymmetries, linking these brain patterns to post-injury return-to-sport outcomes.

However, no studies have yet evaluated the interaction between cortical activation (neural compensations) measured by fMRI and outcomes from targeted neuromotor training during ACL rehabilitation. Understanding brain activation implications is crucial for developing large-scale rehabilitation protocols to reduce the risk of a second, potentially more devastating, knee injury.

This study aims to reveal whether a neuromotor training protocol can positively influence cognitive brain areas related to human movement, particularly by reducing risky injury patterns. It will be the first to test whether dedicated neuromuscular training effectively reduces neural compensations and cortical activation related to non-automated movement, favoring automation areas important for a safe return to sport.

Patients will directly benefit from participating in the innovative neuromotor training program, with functional MRI scans conducted before training begins (post-surgery) and after training completion. Indirectly, the study will assess whether neuromotor training can adapt patient neuromotor patterns to reduce re-injury risk, ultimately benefiting future patients undergoing ACL reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone anterior cruciate ligament reconstruction surgery at any healthcare facility
* Able to understand and consent, adults, who have provided informed consent to participate in the study
* Male or female
* Age between 18 and 30 years at the time of signing the informed consent
* Tegner activity level > 6

Exclusion Criteria:

* History and/or evidence of any neurological disorder or functional impairment;
* Evidence of previous surgeries on the lower limb;
* Inability to provide informed consent;
* Inability to perform the tasks required by the procedure;
* Pregnant or breastfeeding women;
* Oncology patients;
* Contraindications to undergoing MRI examinations.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Variation in the volumetric activation data of the somatosensory cortex | Between 6 and 9 months per patient based on internal analyses and ongoing scientific studies
  Variation in the volumetric activation data of the somatosensory cortex (XYZ coordinates of the peak voxel in non-overlapping brain regions) between timepoint t0 (baseline, pre-training) and timepoint t1 (post-training), measured using fMRI (BOLD sequence). This data allows for the identification of changes in brain activation attributable to the neuromotor training, supporting its effectiveness in reducing neural compensations. Based on the reference literature, a variation equal to or greater than 7 mm in the peak activation coordinates (particularly in the medio-lateral direction) will be considered clinically significant

SECONDARY OUTCOMES:
2D kinematics (in degrees) | Between 6 and 9 months per patient based on internal analyses and ongoing scientific studies
  2D kinematics (in degrees) measured using high-speed cameras on the frontal and sagittal planes, for example, within the 'Green Room' at the Isokinetic Medical Center in Bologna (a room equipped with synthetic turf, high-speed cameras, and an in-floor force platform, used for conducting functional movement tests (15, 26)). These data will allow for the evaluation of the interaction between neural input and biomechanical output following neuromotor training. A variation of at least 5° in key kinematic angles (e.g., knee valgus, lateral trunk tilt) will be considered significant, in accordance with thresholds reported in the literature.
Ground reaction forces | Between 6 and 9 months per patient based on internal analyses and ongoing scientific studies
  Ground reaction forces, measured, for example, using the force platform embedded in the floor of the Isokinetic Green Room. This data will allow evaluation of the interaction between neural input and the force profile exerted on the ground during functional movements. Clinically significant variations will be considered as ≥15% compared to the pre-training value in peak vertical ground reaction force (vGRF, in Newtons) and ≥0.5*BW (force normalized to body weight).
MAT score | Between 6 and 9 months per patient based on internal analyses and ongoing scientific studies
  Movement Analysis Test (MAT) score, calculated based on 2D kinematics and indicative of patient movement quality as recorded, for example, in the 'Green Room' at the Isokinetic Medical Center in Bologna. Specifically, scores of individual sub-criteria (ranging from 0 to 2), which break down movement quality through kinematic thresholds validated in the scientific literature, and the total score (sum of the 5 sub-criteria, ranging from 0 to 10) for each task will be considered. This data will allow evaluation of the interaction between somatosensory cortex activation and a composite index of movement quality across different motor tasks. Any improvement of ≥2 points in the total score (on a 0-10 scale) or ≥1 point improvement in at least three of the five sub-criteria will be considered indicative of significant functional progress, consistent with scientific validation showing a decrease in joint load (dynamic knee valgus moment) as the score increases.
Changes in functional and structural connectivity of brain networks | Between 6 and 9 months per patient based on internal analyses and ongoing scientific studies
  Changes in functional and structural connectivity of brain networks between timepoints t0 (pre-training) and t1 (post-training) assessed using DTI and resting-state (RS) fMRI techniques. A change of ≥0.1 in Fisher z-transformed correlation coefficients between key regions of the motor network (e.g., premotor area, primary motor cortex, SMA) will be considered significant, in accordance with findings reported by Criss et al.
Serious and non-serious adverse events | Between 6 and 9 months per patient based on internal analyses and ongoing scientific studies
  Serious and non-serious adverse events: Most of the events potentially associated with the procedures for outcome collection are expected to be non-serious in nature. Among non-serious adverse events, transient episodes of muscle or joint pain resulting from neuromotor training or perceived fatigue during rehabilitation sessions may occur, without leading to significant clinical consequences. Potentially serious adverse events, although unlikely, could include accidental falls during physical activity causing significant trauma that would require immediate cessation of the procedure and medical intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Ortopedico Rizzoli, Bologna, Italy